CLINICAL TRIAL: NCT04032496
Title: A Randomized Controlled Trial to Investigate a Contemplation-Based Intervention and Health Outcomes in Systemic Lupus Erythematosus Patients
Brief Title: Contemplation-Based Intervention and Health Outcomes RCT in Lupus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, William Cunningham, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 34709
Record Dates: First submitted 2019-06-27; First posted 2019-07-25 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Experimental): Participants in this arm will participate in the Contemplative-Based Intervention for People Living with SLE intervention in addition to one baseline fMRI and blood analysis and one post-treatment fMRI and blood analysis.
  Interventions: Behavioral: Contemplative-Based Intervention for People Living with SLE
- HEP Intervention (Active Comparator): Participants in this arm will participate in the Health Enhancement Program (HEP) intervention in addition to one baseline fMRI and blood analysis and one post-treatment fMRI and blood analysis.
  Interventions: Behavioral: Health Enhancement Program (HEP)

INTERVENTIONS:
Behavioral: Contemplative-Based Intervention for People Living with SLE — Intervention sessions will follow a 6-week format consisting of weekly in-person sessions as well as guided homework to encourage practice at home. Some mindfulness practices that will be included are meditation, group exercise (yoga), group discussions, and deep breathing. Both participants diagnosed with SLE as well as caregivers will participate in the intervention sessions. 5 sessions will be approximately 2 hours long, while the final session will be approximately 4 hours long. Each intervention group will include approximately 4 participants with SLE and 4 caregivers.
  Arms: Mindfulness Intervention
Behavioral: Health Enhancement Program (HEP) — The HEP was designed to create an active control for mindfulness-based stress reduction (MBSR) interventions. The structure of this intervention will mirror that of the other arm of this study, but will lack the mindfulness component. The HEP includes topics such as physical activity, functional movement, music therapy, and nutrition education.
  Arms: HEP Intervention

SUMMARY:
The objective of this study is to test the efficacy of an innovative contemplative-based and caregiver-inclusive intervention can modify pathogenic processes in systemic lupus erythematosus (SLE) compared to a psychoeducation-based intervention. Contemplative techniques such as meditation, mindfulness and yoga may have an impact on the disease burden and may decrease psychological distress, increase self-regulation capabilities, and reduce pain. It is also well documented that social relationships moderate physical health. Incorporating patients' caregivers may strengthen their relationships and thereby improve their health and well-being. It is anticipated that the successful outcome of the mindfulness-based intervention described in this proposal will provide the basis for a new and effective contemplative-based and caregiver-inclusive therapy for SLE and other rheumatic diseases. Although we expect our mindfulness-based intervention to outperform our psychoeducation intervention, we note that the psychoeducation intervention is much closer to treatment as usual (especially insofar as many lupus patients are provided no psychosocial intervention whatever), and to that degree can reasonably be considered our best initial point of comparison. In practice, most patients would be provided medication and some basic information about living with the disease, as well as, perhaps, some additional guidance about coping with chronic stress and pain. We believe that our comparison condition goes beyond this to provide a bona fide intervention in itself.

DETAILED DESCRIPTION:
METHODS: A randomized controlled trial of 50 SLE patients in which subjects receive either a 6-week MBI treatment (n=25) or a 6-week psychoeducation treatment (n=25).

SCREENING: At Visit 1, participants who are deemed eligible for the study will be assigned to either a mindfulness-based intervention group or a psychoeducation intervention group. Participants will also complete the following questionnaires, which will also be administered throughout the intervention schedule:

1. Adverse Childhood Experience (ACE)
2. Adult Attachment Style Questionnaire (AAS; closeness subscale)
3. Brief Health Mindset Scale (BHMS)
4. Center for Epidemiological Studies Depression Scale Revised (CESD-R)
5. Inclusion of Other Self (IOS)
6. Interpersonal Reactivity Index (IRI; empathic concern and perspective-taking subscales)
7. Interpersonal Regulation Questionnaire (IRQ)
8. LupusPRO (patient only)
9. MacArthur Scales of Subjective Social Status (Community and Socioeconomic Status)
10. Caregiver Burden Questionnaire (support person only)
11. Multidimensional Scale of Perceived Social Support (MSPSS)
12. Pain Catastrophizing Scale (PCS)
13. Ruminative Responses Scale (RRS; short form)
14. Social Interaction Phobia Scale (SIPS)
15. State Trait Anxiety Inventory (STAI-T, STAI-S)
16. Ten Item Big Five Questionnaire
17. Toronto Mindfulness Scale (TMS)
18. Lupus Quality of Life
19. CAM Health Belief Questionnaire

INTERVENTIONS: All participants will complete either a 6-week mindfulness-based intervention or a 6-week psychoeducation intervention. All sessions will be in-person in a group setting, and accompanied by homework. For both interventions, participants will practice what they learned on a daily basis as their homework. However, the mindfulness intervention may also have video/audio homework to complete. Sessions 1-5 will last approximately 2 hours each. The final (6th) session will be a retreat that will last approximately 4 hours. Questionnaire data will be collected throughout the intervention.

ASSESSMENTS: Assessment visits 1 and 9 will be performed by rheumatologists and include: complete history, physical examination, information about SLE drug treatment and laboratory examination. Lupus disease activity and damage will be measured by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) and systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI) respectively. Information on socio-demographics, clinical variables (SLEDAI-2K and SDI), co-morbidities (dyslipidemia, atherosclerosis, cerebrovascular disease, and others) are collected as part of the and will be made available for the analysis in this study. Lupus serology (including C3/C4, anti-ds DNA antibodies) and routine blood test (including complete blood count test and chemistry panel) are also collected regularly during the patients' visits to the clinic and will be made available for the analysis in this study.

fMRI Tasks: Participants will complete a series of questionnaires completed within 24 hours after the visit via Qualtrics and a series of tasks while functional MRI data is recorded. After the fMRI, there will be four cognitive tasks done on the computer outside of the scanner. These include:

Continuous Associative Binding (CAB): The goal of this task is to track different aspects of memory and decision-making, in particular the ability of individuals to form associations between pairs of items presented at the same time. In the tasks, participants are presented with pairs of images of objects (e.g., a pencil and a lamp) and their job is to indicate whether the have seen that exact pair of images presented together in the present block of trials.

Flanker: The goal of the flanker task is to measure inhibitory control and decision-making. In each trial, participants are presented with a cluster of arrows pointing either left or right. The task is for the participant to indicate the direction the arrow in the center of the cluster of arrows is pointing.

Random Dot Motion (RDM): The goal of this task is to track attention and perceptual decision-making. In each trial, participants see a circle filled with dots moving in different directions. Most of the dots are moving in random directions, but some of the dots are moving coherently either left or right. The task of the participant is to indicate (either by the keyboard or touch screen) whether more coherent dots are moving to the right or left.

Balloon Analog Risk Task (BART): The goal of this task is to track risk-taking behavior, reinforcement learning, and decision-making. On each trial, the participant indicates whether they would like to pump more air into the balloon, increasing the amount of points/money they could earn if they collect before the balloon pops, or whether they want to collect what they have earned and add it to the bank. If they pump and the balloon pops, they lose the chance to collect that money for that balloon.

Support people will complete a series of questionnaires completed within 24 hours after the visit via Qualtrics and the Handholding Task. The support person is the partner and will be asked to hold hands with the patient for the partner portion of the task. The support person will be connected to the shock device (STM100C Stimulator Module, BIOPAC Systems) for one round of the task, and the shock level will be calibrated to their pain tolerance.

After the fMRI, there will be four cognitive tasks done on the computer outside of the scanner. These include the same tasks for the participant (listed above).

For the scan, standard procedures for removal of all participant ferromagnetic objects (e.g., wristwatches) will be implemented, and the procedures of the study will be reviewed, insuring that participants have an opportunity to ask any remaining questions. All standard fMRI safety screening procedures will be done prior to the fMRI, and female participants will take a urine based pregnancy test. Participants will complete the following tasks while in the scanner:

Resting State Task: Mindfulness training has been shown to alter resting state connectivity in areas related to emotions and stress (e.g., Taren et al., 2015). Thus, we will record resting state data in all visits. Participants will be asked to rest in the scanner. Following the resting state scans, participants will also complete selected questions from the Amsterdam Resting State Questionnaire 2.0 to provide subjective descriptions of their experience.

Hand holding Task: The handholding task is a measure the social regulation of the neural response to threat. Each trial involves the presentation of 12 threat and 12 safety cues in randomized order across blocks of approximately 7 minutes. Participants and partners will be told that threat cues indicate a 17% chance of mild electric shock. These basic threat paradigms will be repeated across 3 blocks of threat/safety cues and counterbalanced across subjects. These blocks will include the alone condition, and the partner hand holding condition in the Threat to Self task, and the partner hand holding condition in the Threat to Partner task. Electric shock will be delivered via an automated computer controlled device (STM100C Stimulator Module, BIOPAC Systems) to the ankle (4 mA, cf., Tursky & O'Connell, 1972). The shock level will be calibrated to each participant's pain tolerance.

Resting State Task (a second time)

All fMRI conditions will be followed by ratings using the Self-Assessment Manikins.

ANALYSIS: The main analysis is planned when all patients have concluded the MBI or psychoeducational program, all data have been entered, verified and validated and the primary database has been locked. Following data reduction and preparation, analysis of all self-report and biological (e.g., fMRI) data will be conducted using hierarchical multilevel modeling procedures designed to maximize sensitivity to both within- and between- subject sources of variation across time, including baseline measurements pre- and post- intervention. In addition to testing for specific group-level effects of intervention, individual differences in response to treatment and/or in biological measures will be assessed as a function of self-report data at both state and trait levels, modeled as interaction effects in multilevel models.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* 18 years of age or older
* Literate in English: able to read, understand, follow instructions, and complete the rating scales and questionnaires accurately
* Have a clinical diagnosis of systemic lupus erythematosus
* Must pass the initial MRI screening
* Must be a participant in The University of Toronto Clinic and Database Research Program - Prognosis and Genetic Studies in Systemic Lupus Erythematosus
* Must be able to access the Internet regularly

Exclusion Criteria:

* Significant previous mindfulness training and experience (e.g. MBSR course, daily meditation practice)
* Any current Axis I DSM-IV-TR psychiatric disorder that, in the clinician's opinion, warrants treatment or would preclude safe participation in the protocol, including, but not limited to: psychosis, schizophrenia, dementia, schizotypal personality disorder, borderline personality disorder, bipolar disorder, primary diagnosis of eating disorder, or chronic suicidality or homicidality.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not related to SLE (i.e., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the treating physician, could confound the results of the study or put the patients at undue risk.
* Chronic use of prescribed or recreational psychoactive drugs (self-reported)
* Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Baseline (self-reported)
* Too sick to meaningfully participate (e.g. hospitalized, flaring at the time of screening)
* In order to participate in the MRI portion of the study, participants must pass the in-person MRI screening administered by the MRI technician before each MRI. If participants fail the in-person MRI screening, they will be excluded from the MRI portion of the study, but can still participate in the intervention portion of the study.
* Is not a participant in The University of Toronto Clinic and Database Research Program - Prognosis and Genetic Studies in Systemic Lupus Erythematosus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in systemic lupus erythematosus (SLE) disease activity | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline SLE Disease Activity Index 2000 (SLEDAI-2K) total score (range from 0 to 105 with higher values representing worse outcomes). Total score represents the sum of the central nervous system, vasculitis, musculoskeletal, renal, skin, serosal, immunologic, fever, and hematologic subscales.

SECONDARY OUTCOMES:
Change from baseline in brain activity during functional MRI | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change in brain activity during functional MRI handholding task
Change from baseline in organ-specific SLE disease activity (central nervous system subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K central nervous system score (range 0-56 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (vasculitis subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K vasculitis score (range 0-8 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (musculoskeletal subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K musculoskeletal score (range 0-8 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (renal subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K renal score (range 0-16 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (skin subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K skin score (range 0-6 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (serosal subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K serosal score (range 0-4 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (immunologic subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K immunologic score (range 0-4 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (fever subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K fever score (range 0-1 with higher values representing worse outcomes).
Change from baseline in organ-specific SLE disease activity (hematologic subscale) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SLEDAI-2K hematologic score (range 0-2 with higher values representing worse outcomes).
Change from baseline in erythrocyte sedimentation rate (ESR) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for ESR (mm/hr)
Change from baseline in antinuclear antibodies (ANA) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for ANA titer
Change from baseline in white blood cell count (WBC), red blood cell count (RBC), platelet levels, and nucleated RBC count | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for WBC, RBC, platelet levels and nucleated RBC count (amount per microliter)
Change from baseline in hemoglobin levels and mean corpuscular hemoglobin concentration (MCHC) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for hemoglobin levels and mean corpuscular hemoglobin concentration (MCHC) (g/dL)
Change from baseline in hematocrit levels, red cell distribution width (RDW), and nucleated red blood cell percentage | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for hematocrit levels, RDW, and nucleated red blood cell percentage (%)
Change from baseline in mean corpuscular volume (MCV) and mean platelet volume (MPV) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for MCV and MPV (fL)
Change from baseline in mean corpuscular hemoglobin (MCH) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for MCH (pg)
Change from baseline in blood sodium, potassium, chloride, carbon dioxide, and anion gap (mmol/L) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for baseline in blood sodium, potassium, chloride, carbon dioxide, and anion gap (mmol/L)
Change from baseline in blood urea nitrogen, creatinine, glucose, and calcium levels | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for blood urea nitrogen, creatinine, glucose, and calcium levels (mg/dL)
Change from baseline in high sensitivity C-reactive protein (CRP) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for CRP (mg/L)
Change from baseline in complement C3 and complement C4 | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for complement C3 and complement C4 (mg/dL)
Change from baseline in cytokine panel (tumor necrosis factor alpha; interleukin 2, 2 receptor (CD25) soluble, 12, gamma, 4, 5, 10, 13, 17, 1 beta, 6, 8) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Abnormal lab values for cytokine panel (pg/mL)
Adult attachment style questionnaire - closeness subscale (AAS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in AAS scores (range from 6-30 with higher scores indicating better outcomes)
Adverse childhood experiences questionnaire (ACE) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in ACE scores (ranging from 0-10 with higher scores suggesting worse outcomes)
Brief Health Mindset Scale (BHMS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in BHMS scores (ranging from 6-36, with higher scores reflecting more adaptive mindsets about health)
Center for Epidemiological Studies Depression Scale (CESD-R) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in CESD-R scores (ranging from 0-80 with higher scores representing worse outcomes. Sum of sadness/dysphoria, loss of interest/anhedonia, appetite, sleep, thinking/concentration, guilt/worthlessness, tired/fatigue, movement/agitation, suicidal ideation subscales).
Inclusion of Other in Self Scale (IOS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in IOS scores (ranging from 1-7 with higher scores representing more relationship closeness)
Interpersonal Reactivity Index (IRI) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in IRI scores (ranging from 0-112 with higher scores indicating higher empathy. Sum of empathic concern, perspective-taking, fantasy, and personal distress subscales).
Interpersonal Regulation Questionnaire (IRQ) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in IRQ scores (ranging from 16-112, with higher scores reflecting better outcomes. Total score is sum of negative-tendency, negative-efficacy, positive-tendency, and positive-efficacy subscales.)
MacArthur Scales of Subjective Social Status (community ladder) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in MacArthur Scales of Subjective Social Status (community ladder score ranging from 1-10 with higher scores indicating better outcomes)
MacArthur Scales of Subjective Social Status (socioeconomic status ladder) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in MacArthur Scales of Subjective Social Status (socioeconomic status ladder score ranging from 1-10 with higher scores indicating better outcomes)
Caregiver Burden Questionnaire (CBQ) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in CBQ scores (ranging from 0-88 with higher scores representing worse outcomes)
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in MSPSS scores (ranging from 12-84 with higher scores indicating better outcomes. Sum of family, friends, and significant other subscales)
Pain Catastrophizing Scale (PCS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in PCS scores (ranging from 0-52 with higher scores representing worse outcomes. Sum of rumination, magnification, and helplessness subscales)
Ruminative Responses Scale (RRS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in RRS scores (ranging from 10-40 with higher scores representing worse outcomes. Sum of brooding and reflection subscales).
Social Interaction Phobia Scale (SIPS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in SIPS scores (ranging from 0-56 with higher scores representing worse outcomes. Sum of social interaction anxiety, fear of overt evaluation, and fear of attracting attention subscales).
State Trait Anxiety Inventory (STAI) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in STAI scores (ranging from 40-160 with higher scores representing worse outcomes. Sum of trait anxiety and state anxiety subscales)
Ten Item Personality Inventory (TIPI) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in TIPI scores on each of conscientiousness, openness to experience, extraversion, agreeableness, and neuroticism personality traits (ranging from 1-7 on each personality trait with higher scores representing more expression of each personality trait.)
Toronto Mindfulness Scale (TMS) | Baseline Assessment within 2 weeks prior to intervention, within 2 weeks after intervention
  Change from baseline in TMS scores (ranging from 0-52 with higher scores representing greater mindfulness. Sum of curiosity and decentering subscales)

CONTACTS AND LOCATIONS:
Overall Officials: William A Cunningham, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No